CLINICAL TRIAL: NCT03952312
Title: Feasibility of OncoTool to Improve Self-Management and Adherence to Oral Anticancer Medications
Brief Title: Oncotool for Cancer Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Betina Yanez, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00207397
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cancer; Cancer, Treatment-Related; Medication Adherence; Communication; Tyrosine Kinase Inhibitor
Keywords: eHealth; Adherence; Symptom Burden; Health Related Quality of Life
MeSH Terms: conditions — Neoplasms; Neoplasms, Second Primary; Medication Adherence; Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "OncoTool" Intervention (Experimental)
  Interventions: Behavioral: Oncotool Intervention (symptom reporting + TKI education)
- "Oncotool" Control (Active Comparator)
  Interventions: Behavioral: Oncotool Control (health information)

INTERVENTIONS:
Behavioral: Oncotool Intervention (symptom reporting + TKI education) — OncoTool is a website intended to improve self-management practices for helping cancer patients cope with side effects and improve health-related quality of life. OncoTool provides symptom education and management for dealing with the numerous physical and mental side effects associated with TKIs (e.g., fatigue, nausea, skin toxicity). OncoTool is a website designed to improve TKI adherence by improving quality of life and TKI associated symptom burden, as well as providing a portal for provider-patient communication via a bi-weekly health questionnaire. Both intervention and active comparator conditions are administered to participants for 8 weeks.
  Arms: "OncoTool" Intervention
Behavioral: Oncotool Control (health information) — OncoTool is a health promotion website with health education on subjects like nutrition and exercise specific to cancer patients, as well as general advice on lifestyle choices and prevention. The Oncotool control has similar TKI education content as the experimental content but without the side effect education or physician notification. Both intervention and active comparator conditions are administered to participants for 8 weeks.
  Arms: "Oncotool" Control

SUMMARY:
The purpose of this study is to examine the efficacy of a psychosocial eHealth intervention on the proposed primary outcomes, TKI adherence and health related quality of life (HRQoL), in patients taking TKIs for cancer management.

The intervention components include psychosocial management strategies, cancer medication knowledge and embedded physician reports. The intervention will be delivered via an online application over an 8-week period. Participants in the intervention will complete bi-weekly side effect questionnaires as part of their study involvement, which may trigger an alert to their prescribing physician if they reach a certain threshold. Participants in the control will not complete these questionnaires.

Participants are randomized into either an intervention application (described above) or a control application (health information and general health promotion strategies). Aside from having access to the online application for the recommended 8 weeks, participation in this study includes three assessments: baseline (at the beginning of the research study), post-intervention (8 weeks after baseline) and a 6-month follow-up.

DETAILED DESCRIPTION:
Molecularly targeted tyrosine kinase inhibitors (TKIs) have improved the overall prognosis of patients with cancer. When properly adhered to, TKIs can extend progression-free survival by decades. Despite the promise of TKIs, nonadherence is problematic and studies report that as little as 23% of patients are fully adherent over time. Poor adherence is of significance as it is associated with disease progression and mortality. Despite the importance of optimal adherence (<90% adherence for TKIs), only a handful of interventions with very limited documented efficacy have targeted adherence to TKIs. This is problematic as the number of patients receiving oral anticancer medications is steadily increasing and patients taking TKIs are required to be adherent for years to impact survival. Furthermore, the limited half-life of TKIs highlights the need to optimize full adherence to these medications.

The few interventions that have sought to improve oral anticancer medication adherence have been limited by: (a) lack of a conceptual model that incorporates modifiable psychosocial factors (e.g., illness perceptions, self-efficacy) known to influence adherence behaviors, (b) lack of patient-centered education and training to manage the chronic and debilitating burden of the medication side effects, and (c) lack of more than one objective method of tracking participants' medication adherence. Strategies that (a) facilitate patient-provider communication about side effects and side effect monitoring, and (b) incorporate evidence-based tools to improve side effect monitoring and management, as well as coping with illness-related stress, may be especially beneficial for aiding patients to optimally adhere to TKI medications. Therefore, the investigators propose that an evidence-based psychosocial intervention that can improve management of oral anticancer medication side effects, and therefore improve quality of life, may also improve adherence.

Previous work elucidating the determinants of adherence to oral anticancer medications and developing web-based symptom monitoring tools and psychosocial interventions for patients with cancer makes the research team uniquely positioned to develop and evaluate the feasibility of an intervention to improve adherence to life-saving TKI medications. Consistent with PA-17-061 (Oral Anticancer Agents), the investigators propose to establish the feasibility of an evidence-based, web-delivered and adaptive program called Oncotool to improve adherence to TKIs. Oncotool is patient centered and grounded in models of health behavior change, self-management and established barriers (e.g., patient, system and treatment factors) to medication adherence. Oncotool will incorporate patient education (e.g., compliance education, medication adherence benefits), track side effects bi-weekly, notify providers of patient-reported side effects, and provide medical and psychosocial management strategies for TKI medication side effects. The purpose of this study is to compare the efficacy of Oncotool to a control program, which will contain general health information such as cancer screening, diet and physical activity. The primary study outcome will be feasibility of Oncotool (i.e., acceptability, demand, practicality). Adherence and health-related quality of life (HRQoL) will be assessed as secondary outcomes over 6 months in Oncotool compared to the control condition.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. medical chart confirmed diagnosis of cancer
3. willingness to be randomized into study
4. have initiated TKIs within the past 18 months, as data in literature indicates that the majority of patients who initiate oral anticancer medications are still adherent within the first few months
5. willing to use a web-based platform on a bi-weekly basis, as well as an email address and access to the internet
6. English speaking, as all material will be in English

Exclusion Criteria:

(a) significant cognitive impairment, inpatient psychiatric treatment, or overt signs of severe psychopathology (e.g., psychosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-08-13 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Change in Self Reported Adherence to TKIs will be evaluated with the ARMS questionnaire. | Time Frame: T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention)
  The ARMS (Adherence to Refills and Medications Scale) survey is a previously validated patient-report measure of barriers to medication adherence and adherence-related behavior.
Electronically Verified TKI Adherence will be measured using medication event monitoring systems (MEMS) | ime Frame: MEMS data will be collected continuously during study participation from T1 (prior to starting intervention) to T3 (6 months post-intervention)
  A MEMS cap is an electronic bottle cap that tracks when participants open their medication bottle. MEMS cap data will be collected continuously during the duration of participation in the study.
Pharmacy reported Adherence to TKIs will be measured using pharmacological records | T3 (6 months post-intervention)
  Pharmacy data will be pulled once at approximately T3 when a participant finishes the study. This data will inform how frequently patients refill their oral cancer medication (TKIs).
Change in Health Related Quality of Life will be evaluated with The Functional Assessment of Cancer Therapy (FACT-G7) | T1 (prior to starting intervention), biweekly during the 8 week intervention, T2 (8 weeks post intervention), T3 (6 months post-intervention)
  The FACT-G7 is a validated questionnaire that assesses top-rated symptoms and concerns for a broad spectrum of advanced cancers.

SECONDARY OUTCOMES:
Cancer-Specific Distress will be evaluated using The Impact of Event Scale (IES) | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention)
  The IES is made up of two subscales measuring the frequency of intrusion and avoidance experiences after a stressful event. The IES has been widely used among patients diagnosed with cancer.
Stress Management Skills will be evaluated with the Brief COPE Inventory | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention)
  The Brief COPE is made up of various subscales measuring different ways of coping. Each question as participants to rate how often they have used each coping mechanism in response to their cancer experience.
Perceived benefits and cost barriers to using oral cancer medications will be assessed using a Beliefs about Medicines scale | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention)
  The 11 point Beliefs about Medicines questionnaire assesses patients' beliefs about the efficacy of their treatment as well as their beliefs about how the benefits and side affects of oral cancer medications affect their life.
Emotional Social Support is assessed using the emotional subscale portion of the Medical Outcomes Study - Social Support Survey Instrument (MOS-SSS) | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention)
  The 8 question MOS-SSS scale was developed by RAND Healthcare to assess the degree of companionship, assistance, or other types of social support that participants have access to. This study will use the 8 question emotional-informational support subsection.
Patient Self-Efficacy in managing side effects is measured using the PROMIS Self Efficacy for Managing Symptoms | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention)
  The PROMIS Self Efficacy for Managing Symptoms survey is a validated, computer adaptive survey to assess how confident participants are in their ability to manage their symptoms and side effects
Cancer Related Communication and Attitudinal Self Efficacy will be evaluated using the Communication and Attitudinal Self-Efficacy scale for cancer (CASE-cancer) | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention)
  The CASE-cancer questionnaire is made up various subscales measuring cancer related communication and attitudinal self-efficacy. Each question asks participants to use a four-point response scale to agree or disagree with statements regarding their level of confidence with different skills.
TKI specific side effects will be evaluated using measures from PRO-CTCAE | T1 (prior to starting intervention), bi-weekly during the 8 week intervention,.T2 (8 weeks post intervention), T3 (6 months post-intervention)
  PRO-CTCAE is a patient-reported outcome measurement system developed by the National Cancer Institute to capture symptomatic adverse events in patients on cancer clinical trials. Measures specific to reported TKI side effects have been chosen for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Betina Yanez, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with any researchers outside Northwestern.

DOCUMENTS (1):
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT03952312/ICF_000.pdf